CLINICAL TRIAL: NCT02886338
Title: Study of the Feasibility of Magnetic Navigated Capsule Endoscope in the Upper Gastrointestinal Tract Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201505067
Record Dates: First submitted 2016-08-17; First posted 2016-09-01 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2016-06

CONDITIONS: Healthy Patient on Good Condition
MeSH Terms: interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsule endoscopy examination (Experimental): Capsule endoscopic examination for the esophagus, stomach and duodenum.
  Interventions: Device: capsule endoscopy

INTERVENTIONS:
Device: capsule endoscopy — The magnetic navigated CE would enable detailed investigations of the whole upper gastrointestinal tract, including the esophagus, stomach and duodenum. Using this remote magnetic manipulation, capsule endoscope might improve diagnostic accuracy and extend the examination of specific area of interest in the gastrointestinal tract.

SUMMARY:
External control of capsule endoscopy (CE) by means of an applied magnetic field is a possible way to maneuver the movement of CE in gastrointestinal (GI) tract. The aim of this study was to evaluate the safety and feasibility of magnetic maneuvering of a capsule endoscope in the upper gastrointestinal tract, including the esophagus, stomach and duodenum in healthy subjects.

DETAILED DESCRIPTION:
Since their introduction in clinical practice in 2000, capsule endoscopy (CE) have widely used as a noninvasive endoscopic examination of the gastrointestinal disorders. Compared with traditional endoscopy, CE has had a significant impact in gastroenterology for diagnoses of gastrointestinal (GI) diseases, largely owing to the following three reasons. First, wireless CE is much more comfortable for the patient. Second, it is much easier and safer to perform. Third, it allows visualization of anatomical regions currently precluded to traditional endoscopy. However, CE does not allow the operator to control the navigation. The movement of the capsule is passive, as it proceeds by means of visceral peristalsis and gravity. This makes the movement of the capsule purely random, so that some portions of the gastrointestinal surface are unable to be visualized. Moreover, if gastrointestinal lesions are identified, the endoscopist cannot maneuver the capsule to perform back and forth, or right and left movement to do further detailed observations. All of these factors contribute to limit the diagnostic values of CE examination.

External controllability of CE by means of an applied magnetic field is a possible solution to the maneuvering problem. However, there is no effective system with straightforward clinical applicability till now. This is ascribable to a lack of reliable magnetic instrumentation suitable for such a purpose. We have reported that using magnetic field navigator can effectively control the locomotion of CE. We have demonstrated, both in vitro and ex vivo, that magnetic field navigator has great potential and practicability of achieving high-precision rotation and controllable movement of CE.

The aim of this study was to evaluate the safety and feasibility of magnetic maneuvering of a capsule endoscope in the upper gastrointestinal tract, including the esophagus, stomach and duodenum in healthy subjects. The movement of the endoscopic capsule in the esophagus could be driven by an external magnetic control device. The external magnetic control device could also adjust the direction of movement of the capsule in the stomach and duodenum, which might make the examination of the whole upper gastrointestinal tract possible. The magnetic navigated CE would enable detailed investigations of the whole upper gastrointestinal tract, including the esophagus, stomach and duodenum. Using this remote magnetic manipulation, capsule endoscope might improve diagnostic accuracy and extend the examination of specific area of interest in the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 adults had experience on insudative upper endoscopy without any contraindication.

Exclusion Criteria:

1. Patient with obstruction of gastrointestinal tract.
2. Pregnant woman.
3. Patient implantation of pacemaker.
4. Patient implanted with metal electronic devices、artificial joints or fixator.
5. Patient with cancer.
6. Patient with difficulty in swallowing.
7. Patient with operation on the stomach.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fat Moon Suk, Study Director — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Capsule Endoscopy Group: The movement of the endoscopic capsule in the esophagus could be driven by an external magnetic control device. The external magnetic control device could also adjust the direction of movement of the capsule in the stomach and duodenum, which might make the examination of the whole upper gastrointestinal tract possible.
  capsule endoscopy: The magnetic navigated capsule endoscope would enable detailed investigations of the whole upper gastrointestinal tract, including the esophagus, stomach and duodenum. Using this remote magnetic manipulation, capsule endoscope might improve diagnostic accuracy and extend the examination of specific area of interest in the gastrointestinal tract.
Period: Overall Study
Arm/Group | Capsule Endoscopy Group
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Capsule Endoscopy Group: Capsule endoscopy group: Participants swallowed a magnetic-assisted capsule endoscope, and an external magnetic field navigator is used for magnetic capsule manipulation in the upper gastrointestinal tract.
  The movement of the magnetic capsule endoscope can be driven by an external magnetic field navigator. The external magnetic field navigator can also adjust the direction of movement of the capsule in the stomach and duodenum. Through the external magnetic-mediated navigation of the capsule in the upper gastrointestinal tract, clinicians can potentially examine the whole upper gastrointestinal tract.
Arm/Group | Capsule Endoscopy Group
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 9

OUTCOME MEASURES:

1. Primary Outcome: Assess the Completeness of Capsule Endoscopy
Description: Evaluate the completeness of capsule endoscopic examination. Visualization of the mucosa of esophagus, stomach and duodenum is analyzed separately during and after the capsule endoscopic examination by real time image and capsule video images. We evaluate the percentage of mucosa that can be clearly examined with a 5-point assessment scale (0%, 25%, 50%, 75% and 100% of the visibility of the mucosa of esophagus, stomach, and duodenum)
Time Frame: The outcome measure was performed within 2 weeks after examination
Population: Subjects had completed the magnetic capsule endoscopic examination
Measure: Mean (Full Range); unit: percentage of mucosa visibility
Arm/Group | Capsule Endoscopy Group
Number analyzed (Participants) | 9
percentage of mucosa visibility
  Percentage of visibility of Mucosa : esophagus | 100 [100 to 100]
  Percentage of visibility of Mucosa: stomach | 85.2 [61.1 to 100]
  Percentage of visibility of Mucosa: duodenum | 86.1 [83.9 to 88.9]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected during the study period for 6 months
Description: No severe adverse event happened in this study. All capsules were successfully retrieved after the capsule endoscopic examination
Groups:
- Healthy Subjects With Capsule Endoscopy Examination: We included participants who were aged from 20 to 65 years. Exclude from the study were those (A) who had obstruction of the GI tract; (B) were pregnant; (C) had pacemaker implantation; (D) were implanted with metal or electronic devices, artificial joints or fixators (E) had cancer; (F) had difficulty in swallowing; (G) had a history of stomach operation.
  All participants received the capsule endoscopic examination for the esophagus, stomach and duodenum.
Arm/Group | Healthy Subjects With Capsule Endoscopy Examination
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes